CLINICAL TRIAL: NCT06630663
Title: Effectiveness of a Wearable Device and AI-Supported Diet and Exercise Intervention in Obese Adults-a Quasi-experimental Design Study
Brief Title: A Wearable Device and AI-Supported Diet and Exercise Intervention
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202011101RINB
Record Dates: First submitted 2024-09-24; First posted 2024-10-08 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-01

CONDITIONS: Obesity and Obesity-related Medical Conditions
Keywords: obesity; weight loss; galactin-1; diet and exercise program
MeSH Terms: conditions — Obesity; Weight Loss | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- standard care (Active Comparator): The standard dietary education encompasses instruction on the calculation of total caloric intake and emphasizes the principles of the Mediterranean diet. Tailored dietary concepts are developed based on individual patient habits to give practical advice. Each participant who chose an extra wearable device downloaded the APP to connect with the health management platform. User interface of the health management platform collected data on the number of steps walked, distance, and heart rate spontaneously. Participants recorded a dietary diary every day with a smartphone APP. All collected information was uploaded to the health management platform, too. The well-trained case managers offered a platform to coach the participants to set-up a better self-managed lifestyle modification through strategies of emphasize reminders, tracking / monitoring/ feedback and goals / rewards.
  Interventions: Behavioral: standard care
- A Wearable Device and AI-Supported Diet and Exercise intervention (Experimental): The standard dietary education encompasses instruction on the calculation of total caloric intake and emphasizes the principles of the Mediterranean diet. Tailored dietary concepts are developed based on individual patient habits to give practical advice. Each participant who chose an extra wearable device downloaded the APP to connect with the health management platform. User interface of the health management platform collected data on the number of steps walked, distance, and heart rate spontaneously. Participants recorded a dietary diary every day with a smartphone APP. All collected information was uploaded to the health management platform, too. The well-trained case managers offered a platform to coach the participants to set-up a better self-managed lifestyle modification through strategies of emphasize reminders, tracking / monitoring/ feedback and goals / rewards.
  Interventions: Behavioral: A Wearable Device and AI-Supported Diet and Exercise intervention

INTERVENTIONS:
Behavioral: A Wearable Device and AI-Supported Diet and Exercise intervention — The standard dietary education encompasses instruction on the calculation of total caloric intake and emphasizes the principles of the Mediterranean diet. Tailored dietary concepts are developed based on individual patient habits to give practical advice. Each participant who chose an extra wearable device downloaded the APP to connect with the health management platform. User interface of the health management platform collected data on the number of steps walked, distance, and heart rate spontaneously. Participants recorded a dietary diary every day with a smartphone APP. All collected information was uploaded to the health management platform, too. The well-trained case managers offered a platform to coach the participants to set-up a better self-managed lifestyle modification through strategies of emphasize reminders, tracking / monitoring/ feedback and goals / rewards.
  Arms: A Wearable Device and AI-Supported Diet and Exercise intervention
Behavioral: standard care — The standard dietary education encompasses instruction on the calculation of total caloric intake and emphasizes the principles of the Mediterranean diet. Tailored dietary concepts are developed based on individual patient habits to give practical advice. Each participant who chose an extra wearable device downloaded the APP to connect with the health management platform. User interface of the health management platform collected data on the number of steps walked, distance, and heart rate spontaneously. Participants recorded a dietary diary every day with a smartphone APP. All collected information was uploaded to the health management platform, too. The well-trained case managers offered a platform to coach the participants to set-up a better self-managed lifestyle modification through strategies of emphasize reminders, tracking / monitoring/ feedback and goals / rewards.
  Arms: standard care

SUMMARY:
This study implemented a personalized 6-month diet and exercise program to promote weight loss. Participants were recruited from outpatient clinics at the Department of Family Medicine, National Taiwan University Hospital. Overweight and obese adults were eligible, defined as follows: overweight (BMI 24-27 kg/m²), mild obesity (BMI 27-30 kg/m²), moderate obesity (BMI 30-35 kg/m²), and severe obesity (BMI ≥ 35 kg/m²). Exclusion criteria included recent weight changes exceeding 3%, a history of bariatric surgery, untreated psychiatric disorders, or medications affecting body weight.

Study design: Of the 171 subjects screened, 29 were excluded due to BMI criteria, leaving 142 participants for baseline body composition and biochemical analysis. Of these, 98 joined the 6-month weight loss program, while 44 remained in the control group. Participants were divided into two groups: one followed a standard diet and exercise program, while the other used a wearable device and AI apps alongside the same program. The wearable device tracked steps, heart rate, and estimated calories burned. Outpatient visits occurred at weeks 0, 12, and 24, with additional diet and exercise education. Phone consultations at weeks 2, 4, and 8 provided 10-minute guidance sessions from case managers. Weight loss medications were not permitted during the study.

Data collection: Weight, height, and blood pressure were measured using standard scales and sphygmomanometers. Waist circumference was measured by a trained operator, and bioelectrical impedance analysis was used to assess skeletal muscle, fat mass, and body fat percentage. Blood samples were collected after an 8-hour fast to measure glucose, cholesterol, and triglycerides. Insulin levels were measured, and HOMA-IR was used to assess insulin resistance. Galectin-1 levels were measured using an ELISA kit. Measurements were taken at baseline and at the end of the intervention (week 24).

Diet and exercise intervention: All participants followed a standard diet and exercise program. Those opting for the wearable device aimed for 7,500 steps per day, following World Health Organization recommendations for 150 minutes of moderate aerobic activity per week. Dietary education included caloric intake calculations and Mediterranean diet principles. Participants using wearable devices logged daily steps and food intake, which was uploaded to a health management platform. Case managers provided lifestyle coaching through the platform.

DETAILED DESCRIPTION:
Introduction The prevalence of obesity has grown globally, and leading to increases in obesity-related conditions and the medical costs of obesity. Obesity is a complex endocrine and metabolic disorder with features of adipose tissue inflammation, remodeling hypertrophy and hyperplasia of adipocytes. Furthermore, obesity induces an imbalance in the regulation of adipokines, which are a group of cytokines that are produced and secreted in adipose tissue. Many studies have investigated the role of different adipokines, and galectin-1 (Gal-1) has emerged as a novel adipokine. Galectins are carbohydrate-binding proteins with an affinity for β-galactosides. Gal-1 is expressed by various tissues and exhibits a wide range of biological activities. Evidence has indicated that galectin-1 is a regulator of immune responses, inflammation, allergy, homeostasis and development.Gal-1 mainly performs an anti-inflammatory role. However, only in recent years have studies shown that the pro-inflammatory properties of Gal-1 in certain diseases, indicating the dual effects of Gal-1.The expression of Gal-1 is highest in subcutaneous adipose tissue. Gal-1 has been proposed as a novel adipokine that circulates during adipocyte differentiation and adipose tissue homeostasis in the literature.In human studies, circulating Gal-1 is positively associated with body mass index (BMI),body fat and waist circumference.

The promotion of physical activity/exercise training and weight loss is advocated to reduce cardiovascular risk in overweight and obese patients. Exercise training programs consistent with the minimum physical activity guidelines are associated with cardiovascular health benefits.With the development of technology, wearable device plus artificial intelligence APPs can be an effective and low-cost tool for patients by helping facilitate their interactions with health care providers. In a systemic review focused on the characteristics of fitness APPs and wearables to assist users overcome obesity and discovered that the wearables emphasize reminders, tracking / monitoring/ feedback and goals / rewards. The use of wearable devices for improving health care processes and outcomes is promising for health promotion among patients with chronic diseases such as obesity and diabetes.

The level of circulating Gal-1 after diet- and exercise-induced body composition changes has previously never been examined. Therefore, we implemented a 6-month diet and exercise program which applied wearable device plus artificial intelligence APPs to investigate the association of changes in circulating Gal-with weight loss, body composition and metabolic parameters among individuals with obesity.

Materials and Methods Participants This study adopted a personalized 6-month personalized diet and exercise program to promote weight loss. Subjects were recruited in outpatient clinics at the Department of Family Medicine, National Taiwan University Hospital. Overweight and obese adults were eligible for this study. The criteria for overweight and obesity in Taiwan are as follows: overweight is defined as 24 ≤ BMI (kg/m2)≤ 27; mild obesity is defined as 27 ≤ BMI (kg/m2) ≤ 30; moderate obesity is defined as 30 ≤ BMI (kg/m2) ≤ 35; and severe obesity is defined as 35 ≤ BMI (kg/m2). The exclusion criteria were as follows: a body weight change greater than 3% in the previous three months; a history of bariatric procedures; untreated psychiatric disorders; or currently using medications known to affect body weight. This study was approved by the Ethics Committee of National Taiwan University Hospital (202011101RINB), and written informed consent was obtained from all participants.

Study design A total of 171 subjects were screened at the outpatient clinics. Twenty-nine of the 171 participants were excluded from the study after screening because their BMI did not meet the criteria. The remaining 142 subjects participated in body composition and biochemical analysis at baseline. Ninety-eight of these subjects were willing to enter the 6-month weight loss program for diet and exercise intervention, while the other 44 subjects preferred to stay in the cohort as the control group. After enrollment, the subjects were divided into two groups based on their preferences: one group participated in a standard diet and exercise program, while the other group received the same program along with a wearable watch and artificial intelligence APPs. The wearable watch could be used to track and monitor various metrics, including steps, heart rates and calorie expenditure. Outpatient clinic visits were scheduled in week 0, week 12, and week 24. Face-to-face diet and exercise education were conducted at each visit. Participants also completed phone consultations in week 2, week 4, and week 8 by the case managers. The case managers provided diet and exercise consultation and coaching for 10 minutes per consultation. Medication for weight loss was not allowed during the training program.

Data collection Participants' weight, height, systolic blood pressure (BP), and diastolic BP were measured by a standard electronic scale of stadiometer and sphygmomanometer. Body weight was assessed to the nearest 0.1 kg with the participant clothed in lightweight clothing. Waist circumference was measured by the same trained operator. Bioelectrical impedance analysis was performed for skeletal muscle, fat-free mass, body fat mass and body fat percentage. Regarding blood analysis, venous blood samples were collected from the participants following a minimum eight-hour fasting period. Serum glucose, total cholesterol, high-density lipoprotein (HDL) cholesterol, low-density lipoprotein (LDL) cholesterol, and triglyceride levels were assessed by an automatic spectrophotometric assay (HITACHI 7250, Japan). Fasting insulin levels were measured by a microparticle enzyme immunoassay using an AxSYM system (Abbott Laboratories, Dainabot Co, Tokyo, Japan). The homeostatic model assessment of insulin resistance (HOMA-IR) was applied as an indirect measure of the degree of insulin resistance (HOMA-IR=fasting insulin x fasting plasma glucose/22.5, with glucose in mmol/L and insulin in mU/L).Serum galectin-1 (cat no: DGAL10, RD Systems, MN, USA) levels were measured by an enzyme-linked immunosorbent assay (ELISA) kit that employed the quantitative sandwich enzyme immunoassay technique. All body composition, blood pressure, and biochemical variables were measured on day 1 (baseline) and at the end of the intervention (week 24).

Diet and exercise intervention The subjects were divided into two groups based on their preferences. Each participant received a standard diet and exercise program. For those who opted for additional wearable devices, a wearable watch and artificial intelligence apps were administered. Each participant was suggested to aim for a daily target of 7,500 steps. This recommendation aligns with the guideline of achieving approximately 150 minutes of moderate-intensity aerobic physical activity per week, as recommended by the World Health Organization.The standard dietary education encompasses instruction on the calculation of total caloric intake and emphasizes the principles of the Mediterranean diet. Tailored dietary concepts are developed based on individual patient habits to give practical advice. Each participant who chose an extra wearable device downloaded the APP to connect with the health management platform. User interface of the health management platform collected data on the number of steps walked, distance, and heart rate spontaneously. Participants recorded a dietary diary every day with a smartphone APP. All collected information was uploaded to the health management platform, too. The well-trained case managers offered a platform to coach the participants to set-up a better self-managed lifestyle modification through strategies of emphasize reminders, tracking / monitoring/ feedback and goals / rewards.

ELIGIBILITY:
Inclusion Criteria:

1. At least 20 years of age
2. BMI ≥24 kg/m2 plus one or more obesity-related comorbidities such as hypertension, diabetes, hyperlipidemia, sleep apnea syndrome, or nonalcoholic fatty liver disease
3. Able to use a wearable device and an app
4. Able to sign the informed consent form after receiving a detailed explanation of the study

Exclusion Criteria:

1. Unable to finish the self-administered questionnaires
2. Unable to complete body composition assessment (bioimpedance analysis and abdominal echo), hand grip test, and blood sampling
3. Unable to return to our clinics at the scheduled time

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-07-10 (Estimated); Primary Completion 2026-01-10 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
weight change | 24 weeks
  The weight change in kilograms from baseline to week 24

SECONDARY OUTCOMES:
waist change | 24 weeks
  The waist change in cm from baseline to week 24
Changes of the serum fasting glucose | 24 weeks
  Changes of the serum fasting glucose in mg/dl from baseline to week 24
Changes of the serum high-density lipoprotein cholesterol | 24 weeks
  Changes of the serum high-density lipoprotein choleste in mg/dl from baseline to week 24
Changes of the low-density lipoprotein cholesterol | 24 weeks
  Changes of the low-density lipoprotein cholesterol in mg/dl from baseline to week24
Changes of the triglyceride | 24 weeks
  Changes of the triglyceride in mg/dl from baseline to week24
Changes of the blood pressure | 24 weeks
  Changes of the systolic and diastolic blood pressure in mmHg from baseline to week24
BMI changes | 24 weeks
  Changes of BMI with weight in kilograms, height in meters from baseline to week24

CONTACTS AND LOCATIONS:
Overall Officials: CW LU, A.P., Study Director — National Taiwan University Hosital
Locations (1):
- National Taiwan University Hospital, Taipei, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No